CLINICAL TRIAL: NCT06233591
Title: A Multicenter, Dose-Ranging Trial Evaluating the Safety, Tolerability, and Efficacy of LP-10 in Subjects With Symptomatic Oral Lichen Planus
Brief Title: Evaluating LP-10 in Subjects With OLP
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Lipella Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 310-001
Record Dates: First submitted 2023-12-19; First posted 2024-01-31 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2024-07

CONDITIONS: Oral Lichen Planus
Keywords: OLP
MeSH Terms: conditions — Lichen Planus, Oral

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- LP-10 0.25mg (Experimental): 0.25mg LP-10 / 10 mL twice daily oral rinse
  Interventions: Drug: LP-10 (Liposomal Tacrolimus)
- LP-10 0.5 mg (Experimental): 0.5mg LP-10 / 10 mL twice daily oral rinse
  Interventions: Drug: LP-10 (Liposomal Tacrolimus)
- LP-10 1.0 mg (Experimental): 1.0mg LP-10 / 10 mL twice daily oral rinse
  Interventions: Drug: LP-10 (Liposomal Tacrolimus)

INTERVENTIONS:
Drug: LP-10 (Liposomal Tacrolimus) — Liposomal oral rinse formulation of Tacrolimus

SUMMARY:
This is a multicenter, dose-ranging study including adult male and female subjects (>= 18 years old) with symptomatic Oral Lichen Planus (OLP). A total of approximately 24 subjects will be enrolled at approximately eight (8) study sites in the United States. This study will evaluate the safety, tolerability and efficacy of LP-10 at 0.25 mg, 0.5 mg and 1.0 mg of tacrolimus.The study consists of screening, treatment and follow-up phases. The treatment phase includes 10 mL LP-10 oral rinse for 3 minutes twice a day for 4 weeks. The follow-up phase includes one post-treatment visit 2 weeks after the last oral LP-10 dose.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent
* Male or female ≥ 18 years of age
* Oral biopsy performed within the last 10 years before the Screening Visit demonstrating OLP and/or oral lichenoid mucositis in the absence of cancer or dysplasia
* Moderate OLP based on an OLP Investigator Global Assessment (IGA) score of ≥ 3
* OLP Pain and Sensitivity Numerical Rating Scale (NRS) score of ≥ 3
* Patients taking prescription oral steroid or rinse treatment(s) at the time of the Screening Visit agree to stop treatment for the duration of the trial and to undergo a 4-week washout period
* Willing and capable of understanding and complying with all requirements of the protocol, including proper completion of the self-administered questionnaires
* Willing to avoid live vaccines while enrolled in the trial
* Patients of child-bearing potential must have a negative pregnancy test and agree to undergo pregnancy testing at each study visit. (unless patient has undergone a bilateral tubal ligation or hysterectomy and/or is post-menopausal as defined by the absence of menses for at least 12 months)
* Patients of child-bearing potential and male participants with a female partner of child-bearing potential, agree to use a reliable method of contraception (condoms and/or oral contraceptives) for the duration of the trial and for 10 days thereafter

Exclusion Criteria:

* Hyperkalemia
* Chronic kidney disease
* Long QT syndrome
* History of oral cavity or oropharyngeal cancers
* Active cancer
* Uncontrolled hypertension (i.e., > 145 mm/Hg systolic or > 95 mmHg diastolic)
* Patients who failed tacrolimus treatment for OLP in the past
* Patient who is currently or has previously participated in another oral cavity therapeutic or device study within 3 months of screening and has not returned to baseline
* History of oral cavity infection (bacterial, viral or fungal) within 3 months prior to screening
* Pregnant or lactating
* Active bleeding peptic ulcer disease
* Known allergy to liposomes and/or egg yolk and/or tacrolimus
* Evidence of renal impairment (creatinine > 2 × the upper limit of normal at Visit 1), hepatic impairment (AST or ALT > 3 × the upper limit of normal at Visit 1), clinically significant cardiovascular, respiratory, or psychiatric diseases per investigator's judgment
* Patients currently taking magnesium and aluminum-hydroxide antacids or metoclopramide
* Patients currently taking aminoglycosides, ganciclovir, amphotericin B, cisplatin, nucleotide reverse transcriptase inhibitors, and protease inhibitors
* The presence of any clinically significant systemic disease or condition that in the opinion of the investigator would make the patient unsuitable for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety of LP-10 in patients with oral lichen Planus | over 4 weeks of treatment and 2 weeks of follow-up
  Incidence and severity of treatment-emergent adverse events, changes in standard laboratory studies, whole-blood tacrolimus levels

SECONDARY OUTCOMES:
To evaluate the preliminary efficacy of LP-10 in patients with oral lichen planus | from baseline to 1 and 4 weeks after the first dose and 2 weeks after the last dose
  Change in the OLP Investigator Global Assessment (IGA) score
To evaluate the preliminary efficacy of LP-10 in patients with oral lichen planus | from baseline to 1 and 4 weeks after the first dose and 2 weeks after the last dose
  Change in the OLP Reticulation, Erythema, and Ulceration (REU) score
To evaluate the preliminary efficacy of LP-10 in patients with oral lichen planus | from baseline to 1 and 4 weeks after the first dose and 2 weeks after the last dose
  Changes in the Oral Lichen Planus Symptom Severity Measure (OLPSSM) score
To evaluate the preliminary efficacy of LP-10 in patients with oral lichen planus | from baseline to 1 and 4 weeks after the first dose and 2 weeks after the last dose
  Change in the OLP Pain and Sensitivity Numerical Rating Scale (NRS)
To evaluate the preliminary efficacy of LP-10 in patients with oral lichen planus | at 4 weeks after first dose
  Patient Global Response Assessment (GRA)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Center for Dermatology, Fremont, California
  - UCSF School of Dentistry, San Francisco, California
  - Miami Cancer Institue at Baptist Health, Inc, Miami, Florida
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Erie County Medical Center, Buffalo, New York
  - Atrium Health Oral Medicine & Maxillofacial Surgery, Charlotte, North Carolina
  - Paddington Testing Co, Inc, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brennan MT, Frustino J, Al-Eryani K, Sroussi H, Parish JL, Routh HB, Dhawan S, Klein GL, Chancellor MB, Villa A. Safety and Efficacy of LP-10 Liposomal Tacrolimus in Oral Lichen Planus: A Multicenter Phase 2 Trial. Dermatol Ther (Heidelb). 2025 Oct 31. doi: 10.1007/s13555-025-01572-2. Online ahead of print. PMID 41174333